CLINICAL TRIAL: NCT01674855
Title: Randomized, Open, Multi-Center, Phase III Study to Evaluate Efficacy and Safety in Chemotherapy-induced Neutropenia of Once-per-cycle DA-3031(PEG-G-CSF) and Daily G-CSF in Patients With Malignancies Receiving Myelosuppressive Chemotherapy
Brief Title: Phase III Study of DA-3031(PEG-G-CSF) in Chemotherapy-induced Neutropenia
Acronym: PEG-G-CSF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA3031_NP_III
Record Dates: First submitted 2012-01-19; First posted 2012-08-29 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Chemotherapy Induced Neutropenia
Keywords: PEG-G-CSF
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor, human; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-3031 (Experimental): PEG-G-CSF
  Interventions: Drug: PEG-G-CSF
- Leucostim® (Active Comparator): G-CSF
  Interventions: Drug: G-CSF

INTERVENTIONS:
Drug: PEG-G-CSF — Prefilled syringe, 6mg/day, single dosing per cycle, for 6 cycle
  Other Names: DA-3031
  Arms: DA-3031
Drug: G-CSF — Vial, 100ug/m2/day, multiple dosing per cycle(daily administration, up to 10 days), for 6 cycle
  Other Names: Leucostim®
  Arms: Leucostim®

SUMMARY:
This study is to determine whether once-per-cycle DA-3031(PEG-G-CSF) is not inferior to daily G-CSF in chemotherapy-induced neutropenia.

DETAILED DESCRIPTION:
Eligible subjects are randomly assigned to receive once-per-cycle DA-3031(PEG-G-CSF) or daily G-CSF(up to 10 days). This study is conducted for 6 cycles of chemotherapy, that each cycle is repeated every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age : ≥18, ≤70
2. Diagnosis of stage II, III or IV breast cancer
3. ANC≥1,500/mm3, Platelet≥100,000/mm3, ECOG : 0 or 1
4. Creatinine < 1.5 x ULN
5. Total bilirubin/AST/ALT < 1.5 x ULN, ALP < 2.5 x ULN
6. Have given a written, informed consent

Exclusion Criteria:

1. Prior chemotherapy
2. Prior bone marrow or stem cell transplantation
3. Other malignancy history within 5 years
4. Prior exposure to pegfilgrastim or filgrastim or other colony-stimulating factors
5. Received any other investigational drugs within 30 days of informed consent date
6. Radiation therapy within 4 weeks of informed consent date
7. Infective symptom before chemotherapy into this study
8. Received systemic antibiotics within 72 hours of randomization into this study.
9. HIV positive
10. Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Duration of grade 4 neutropenia in cycle 1 | 21 day
  Grade 4 neutropenia means the ANC count is less than 500/mm3.

SECONDARY OUTCOMES:
ANC nadir in cycle 1 | 21 day
  ANC nadir means the lowest point of ANC count.
Time to ANC recovery in cycle 1 | 21 day
  ANC recovery means the ANC count is more than 2,000/mm3.
Incidence of febrile neutropenia | 126 day
  Febrile neutropenia means the ANC count is less than 1,000/mm3 and body temperature is more than 38.3 degrees celsius.
Incidence of IV antibiotics administration | 126 day
  IV antibiotics administration means that antibiotics are administered through intravenous route.

CONTACTS AND LOCATIONS:
Overall Officials: JaeHong Seo, M.D., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University GURO hospital, Seoul, South Korea